CLINICAL TRIAL: NCT04295057
Title: Register on the Study of Prevalence and Incidence, Risk Factors and Outcomes of Hospitalizations in Older Age Groups in Eurasia.
Brief Title: Register of Therapeutical Patients Over 60 Years
Acronym: ASCLEPIUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eurasian Association of Therapists (Other)
Responsible Party: Principal Investigator, Tamara Kriukova, Eurasian Association of Therapists, Eurasian Association of Therapists
Other Study IDs: EUAT; ASCLEPIUS (Registry Identifier: ASCLEPIUS)
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Men; Age Problem; Therapeutic Alliance
Keywords: register; therapy
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-intervention — Non-intervention

SUMMARY:
Register for the study of the prevalence and burden of diseases, risk factors and outcomes of hospitalizations in older age groups in the countries of Eurasia.

DETAILED DESCRIPTION:
An open, multicenter registry to track all major noncommunicable diseases and risk factors in older age groups, prescribed drugs, and disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* over 60 years
* Appointment to a doctor of a therapeutic profile

Exclusion Criteria:

* Reluctance of the Patient to participate in the Register;
* Age under 60 at the time of inclusion in the Register.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anonymous men and women in the age group over 60 see a doctor for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence | 12 months
  Incidence of non-infectious diseases
Non-infectious diseases | 12 months
  Age-related non-infectious diseases dynamics of the development of the main after 60 years
Age groups | 12 months
  The prevalence of various non-infectious diseases in different age groups
Therapy | 12 months
  Names, doses and duration of prescribed therapy
Drugs | 12 months
  Analysis of prescribed therapy and calculation of losses from improper treatment due to repeated hospitalizations, disability and complications
Measure criteria | 12 months
  12000 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Eurasian Association of Therapists, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No